CLINICAL TRIAL: NCT03802318
Title: A Comparison Study of Helicobacter Pylori Eradication Rates Between Daily Four Times and Daily Two Times Usage of Proton Pump Inhibitor and Amoxicillin for the First Line and the Second Line Eradication Therapy
Brief Title: Daily Four Times or Two Times Usage of PPI and Amoxicillin for the First or Second Line H. Pylori Eradication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chen, chief, division of hepato-gastroenterology, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201801792A3
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Gastritis; Helicobacter-Associated Pyloric Ulcer
Keywords: Helicobacter pylori; Proton pump inhibitor; Amoxicillin; Urea breath test; Levofloxacin; Clarithromycin
MeSH Terms: interventions — Rabeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HDDT group (Experimental): high dose PPI induction (oral rabeprazole 20mg qid) for 3 days, then 14 days combined with amoxicillin (regular dose, daily 2 g, 500mg qid) for high frequency dual therapy.
  Interventions: Drug: Rabeprazole
- CATT group (Placebo Comparator): conventional triple therapy 14 days (rabeprazole 20 mg bid, amoxicillin 1 g bid, clarithromycin 500 mg bid)
  Interventions: Drug: Rabeprazole
- LHDT group (Experimental): high dose PPI (oral rabeprazole 20mg qid) induction for 3 days, then Rabeprazole 20 mg qid, amoxicillin 500 mg qid, levofloxacin 500 mg qd for 14 days.
  Interventions: Drug: Rabeprazole
- LATT group (Placebo Comparator): levofloxacin base rescue therapy 14 days (rabeprazole 20 mg bid, amoxicillin 1 g bid, levofloxacin 500 mg qd)
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole daily four time (Bid) or daily four times (Qid) Amoxicillin used daily two times (1000 mg bid) or daily four times (500 mg qid) apply in the first line or the second line H pylori eradication therapy
  Other Names: Amoxicillin

SUMMARY:
The hypothesis and plan of the current study are:

1. One induction phase of high dose PPI before eradication will increase intragastric pH and induce H. pylori into an active replicative status. Active replicative status will enhance the bactericidal effect of amoxicillin. Rabeprazole (20 mg) four times per day (qid) for 3 days will be used for induction in this study.
2. High dose PPI will provide adequate plasma concentration irrespective of the CYP2C19 genotype of the population. Here rabeprazole (20 mg) qid will be applied as high dose PPI.
3. High frequent amoxicillin usage (500 mg, qid) will maintain plasma concentration above the MIC. Amoxicillin (500 mg) qid will be described for total 14 days.
4. In the rescue therapy, add levofloxacin on high dose dual therapy will increase the eradication rate than single high dose dual therapy. A combination of levofloxacin and high dose dual therapy will also have a better eradication rate than the common used levofloxacin based triple therapy.

DETAILED DESCRIPTION:
This study aims to evaluate:

1. the first line H. pylori eradication rate of high dose dual therapy with 14 days rabeprazole 20 mg qid, plus amoxicillin 500 mg qid (HDDT group) comparing to the clarithromycin-based triple therapy with 14 days clarithromycin 500 mg bid, amoxicillin 1000mg bid , and rabeprazole 20mg bid (CATT group).
2. the eradication efficacy in rescue therapy of a levofloxacin-based triple therapy with 14 days levofloxacin 500 mg qd, amoxicillin 500 mg qid and rabeprazole 20 mg qid (LHDT group) comparing to the common levofloxacin-based triple therapy with 14 days levofloxacin 500 mg qd, amoxicillin 1000mg bid and rabeprazole 20 mg (LATT group).

Material and Methods Patients and study design This is a prospective, randomized, open-label trial. The patients diagnosed with H. pylori infection will be enrolled from Jan 2019 to Dec 2020 in Keelung Chang-Gung Memorial hospital. The source of subjects may include (1) community participants who obtain a positive result of urea breath test (UBT) from the checkup screening (2) hospital patients who obtain a positive result of H. pylori infection by esophagogastroduodenoscopy (EGD). Exclusion criteria include age less than 20 years, pregnancy or nursing, serious concomitant illness, malignant tumors, history of hypersensitivity to study drugs, active ulcer bleeding, previous gastric surgeries, and taking PPIs within two weeks or antibiotics within one month before study. Patients without previous H. pylori eradication therapy are invited to receive the first-line regimens, whereas patients who have previously received H. pylori eradication therapy are invited to receive rescue regimens.

Hospital patients are asked to receive five endoscopic biopsy specimens (3 from gastric antrum and 2 from body mucosa) for rapid urease test (RUT) and culture studies. The definition of H. pylori infection is a positive finding from UBT, RUT or culture.

Diagnosis for H. pylori infection RUT Three specimens from endoscopic biopsy are used for the RUT (HelicotecUT ® plus test; Strong Biotech Corporation, Taipei, Taiwan). The test result will be read one hour later. A medium color change from yellowish to pink or red is recorded as a positive finding for H. pylori.

Bacterial culture and antibiotic susceptibility test Two specimens are homogenized and streaked onto an agar plate with selective medium. The plates are incubated at 37∘C under microaerophilic conditions (5% O2, 10% CO2, 85% N2) for 3-7 days. H pylori is identified by its characteristic biotyping. The primary isolates are subcultured for antibiotic susceptibility tests as described previously [21]. The E test strips (AB Biodisk, Solna, Sweden) are used for susceptibility testing. The resistance to antibiotics is according to MIC values of >0.5, ≥1, ≥8, and >1 mg/L for amoxicillin, clarithromycin, tetracycline, and levofloxacin, respectively [21].

Subjects should complete a standardized questionnaire and recorded symptoms and daily drug consumption during the treatment period to evaluate compliance and tolerability.

All patients are asked to describe any adverse event (diarrhea, taste disturbance, nausea ⁄ vomiting, bloating, abdominal pain, constipation, headache and skin rash) during the period when they are taking eradication drugs. The incidence of side effects is checked using a standardized degree of interference with daily activities format, as follows: absent; mild-not interfering; moderate-frequently interfering, but allowing treatment to be completed; severe-requiring interruption of treatment [33].

Four weeks after treatment completion, H pylori eradication success will be determined by 13C-UBT.

ELIGIBILITY:
Inclusion Criteria:

* The source of subjects may include (1) community participants who obtain a positive result of urea breath test (UBT) from the checkup screening (2) hospital patients who obtain a positive result of H. pylori infection by esophagogastroduodenoscopy (EGD).

Exclusion Criteria:

* Exclusion criteria include age less than 20 years, pregnancy or nursing, serious concomitant illness, malignant tumors, history of hypersensitivity to study drugs, active ulcer bleeding, previous gastric surgeries, and taking PPIs within two weeks or antibiotics within one month before study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 2~3 months
  Two to three months after eradication therapy, urea breath test will be performed. If the result of UBT is negative, it means successful eradication. If the result is positive, it means eradicaiton failure

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jui Hung, PhD, Study Chair — Chang-Gung Memorial Hospital at Keelung
Locations (1):
- Chang-Gung memorial hospital at Keelung, Keelung, Taiwan